CLINICAL TRIAL: NCT06582836
Title: A Comparative Assessment of Post Extraction Pain in Orthodontic Patients to Evaluate the Effects of Early Engagement of Tooth with Orthodontic Wires. a Single Center Randomized Clinical Trial (RCT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Meenaz Karim, Dr., Universiti Sains Malaysia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: BDC/R/101/19
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Orthodontic Extraction; Orthodontic Treatment; Orthodontic Treatment Via Premolar Extraction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- investigate the effect of prior engagement of tooth with orthodontic appliance on post extraction pa (Experimental): In this randomized clinical trial, 44 patients were recruited who needed bilateral extractions of first premolars in upper arches. Patients were divided into two groups based on the timing of extractions. Group A needed extractions before alignment while Group B needed extractions for retraction of anterior teeth. Group A was sent for extractions first while Group B went for orthodontic bonding and banding procedures for orthodontic treatment. After series of aligning wires (0.014, 0.016, 17x25, 19x25 Heat activated NiTi and 19x25 SS) patients from group B were sent for extractions. For pain assessment, an 11-point numerical rating scale (NRS) were given to record pain intensity at 2, 4, 8, 12 and then 24 hours after extraction for the next 7 days.
  Interventions: Behavioral: The objective of the study was to investigate the effect of prior engagement of tooth with orthodontic appliance on post extraction pain among orthodontic patients

INTERVENTIONS:
Behavioral: The objective of the study was to investigate the effect of prior engagement of tooth with orthodontic appliance on post extraction pain among orthodontic patients — In this randomized clinical trial, 44 patients were recruited who needed bilateral extractions of first premolars in upper arches. Patients were divided into two groups based on the timing of extractions. Group A needed extractions before alignment while Group B needed extractions for retraction of anterior teeth. Group A was sent for extractions first while Group B went for orthodontic bonding and banding procedures for orthodontic treatment. After series of aligning wires (0.014, 0.016, 17x25, 19x25 Heat activated NiTi and 19x25 SS) patients from group B were sent for extractions. For pain assessment, an 11-point numerical rating scale (NRS) were given to record pain intensity at 2, 4, 8, 12 and then 24 hours after extraction for the next 7 days.

SUMMARY:
The goal of this clinical trial is to determine if the timing of tooth extractions (before or after initial orthodontic treatment) affects pain levels in patients who need bilateral extractions of first premolars in the upper jaw. The participants in this study are patients who require these extractions as part of their orthodontic treatment.

The main questions it aims to answer are:

1. Does extracting teeth before starting orthodontic treatment result in different pain levels compared to extracting teeth after alignment?
2. How do pain levels change over time after the extractions in each group?

Researchers will compare Group A (patients who have extractions before orthodontic treatment) to Group B (patients who have extractions after initial alignment) to see if the timing of the extractions affects pain levels.

Participants will:

Undergo tooth extractions either before or after initial alignment based on their group.

Rate their pain on an 11-point numerical rating scale at various times (2, 4, 8, 12, and 24 hours after extraction, and then daily for a week).

ELIGIBILITY:
Inclusion Criteria:

* 12 to 18-year-old orthodontic patients needing bilaterally symmetrical extractions of first premolars as a part of orthodontic treatment. Angles class I with moderate to severe crowding cases, bimaxillary proclination, and Angles class II division 1 were included.

Exclusion Criteria:

* Patients with poor oral hygiene, carious or missing premolars, multiple missing teeth, systemic diseases, periodontitis or patients on analgesics (NSAIDs, and corticosteroids) were excluded from the study.

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 44 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
A comparative assessment of post extraction pain in orthodontic patients to evaluate the effects of early engagement of tooth with orthodontic wires. | 2.6 years
  In this randomized clinical trial, 44 patients were recruited who needed bilateral extractions of first premolars in upper arches. Patients were divided into two groups based on the timing of extractions. Group A needed extractions before alignment while Group B needed extractions for retraction of anterior teeth. Group A was sent for extractions first while Group B went for orthodontic bonding and banding procedures for orthodontic treatment. After series of aligning wires (0.014, 0.016, 17x25, 19x25 Heat activated NiTi and 19x25 SS) patients from group B were sent for extractions. For pain assessment, an 11-point numerical rating scale (NRS) were given to record pain intensity at 2, 4, 8, 12 and then 24 hours after extraction for the next 7 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Baqai Medical University, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided